CLINICAL TRIAL: NCT04195711
Title: Comparative Validation of the Birefringent Amblyopia Screener With Isolated Small-angle Strabismus
Brief Title: Comparative Validation of "Blinq" and "2WIN" Vision Screeners
Status: Completed | Type: Observational
Sponsor: Alaska Blind Child Discovery (Other)
Responsible Party: Sponsor
Other Study IDs: ABCD blinq 2WIN
Record Dates: First submitted 2019-11-28; First posted 2019-12-12 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2019-12

CONDITIONS: Strabismic Amblyopia; Refractive Amblyopia; Strabismus
Keywords: vision screening, amblyopia
MeSH Terms: conditions — Amblyopia; Strabismus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- blinq screened: Patients screened by new birefringent screener
  Interventions: Diagnostic Test: objective pediatric vision screen, "blinq,"

INTERVENTIONS:
Diagnostic Test: objective pediatric vision screen, "blinq," — hand-held birefringent screener for simultaneous foveation
  Other Names: photoscreen, birefringent screen

SUMMARY:
After 28 years of development, the binocular birefringence screener ("blinq," "Rebion") was commercially released. It need to be validated with AAPOS (American Association for Pediatric Ophthalmology and Strabismus) criteria in part because the next Uniform Standards document is pending.

Adult and children pediatric and strabismus patients were screened with blinq and "2WIN" photoscreener with "CR" corneal reflex alignment test and then compared to confirmatory exam with age-appropriate determination of binocular status.

DETAILED DESCRIPTION:
As a part of a new or follow-up comprehensive eye examinations, patients were screened with two novel objective devices according to AAPOS Uniform guidelines. Following the refractive, alignment and sensory testing, cycloplegic refraction was performed 30 or more minutes after cyclopentolate 1% drops. In cooperative patients, sensory tests including Worth 4-dot, Stereo Fly and "PDI Check" were performed to characterize binocularity. For younger patients, binocular function was estimated by Bruckner Test, 4- base out prism cover and the CR corneal reflex component of "2WIN" photoscreener ("Adaptica," Padova Italy).

Each patient was screened with a recently commercially released blinq screener according to manufacturer's recommendations. If an initial interpretation of "pass" or "refer" was not achieved, then repeat efforts with "timed out" or "inconclusive" were accomplished and results evaluated as if a "refer." An example of blinq birefringent screening is shown in [video].

Patients were screened with the binocular infrared autorefractor "2WIN" according to manufacturer guidelines. Refractive referral criteria were not age-stratified.

The "Rebion blinq" is a unique screening method and therefore we sought to provide appropriate validation. In addition to non-age stratified AAPOS 2003 Uniform guidelines, we collected all cases characterized by constant or persistent strabismus whether large- or small angle employing cover test, 4 base out test, Bruckner Test and "2WIN CR" function. We did not employ any method of retinal videographic analysis of fixation instability.

De-identified patient data recorded for sharing on study website.

ELIGIBILITY:
Inclusion Criteria:

Children in Pediatric Ophthalmology Practice Adult strabismus patients

-

Exclusion Criteria:

patients with enucleations patients with eviscerations patients with exenterations

-

Ages: 1 Year to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients in pediatric eye and adult strabismus practice
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
2003 AAPOS Uniform Amblyopia Risk Factor (ARF) Prevalence | 1 week
  presence of refractive risk factor (anisometropia >1.5 D, hyperopia>3.5 D, astigmatism ≥1.5 D, myopia 3 D or more) and/or strabismus constant >10 PD

SECONDARY OUTCOMES:
Binocularity | 1 week
  Any defective Sensory (stereopsis > 200 sec arc, ocular Worth 4-Dot suppression distance and/or near) and/or objective ocular alignment (positive Bruckner Test, positive 4 prism base out test, or "2WIN" "CR" corneal reflex alignment > 10 PD)

CONTACTS AND LOCATIONS:
Locations (1):
- Alaska Children's EYE & Strabismus, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: Yes
de-identified via website
Supporting Information: CSR
Time Frame: 1 month from now, ongoing
Access Criteria: Study website
URL: http://www.abcd-vision.org/references/index.html

REFERENCES:
- [Background] Birch EE, Subramanian V, Weakley DR. Fixation instability in anisometropic children with reduced stereopsis. J AAPOS. 2013 Jun;17(3):287-90. doi: 10.1016/j.jaapos.2013.03.011. PMID 23791411
- [Background] Gramatikov BI, Irsch K, Wu YK, Guyton DL. New pediatric vision screener, part II: electronics, software, signal processing and validation. Biomed Eng Online. 2016 Feb 4;15:15. doi: 10.1186/s12938-016-0128-7. PMID 26847626
- [Background] Arnold SL, Arnold AW, Sprano JH, Arnold RW. Performance of the 2WIN Photoscreener With "CR" Strabismus Estimation in High-Risk Patients. Am J Ophthalmol. 2019 Nov;207:195-203. doi: 10.1016/j.ajo.2019.04.016. Epub 2019 May 9. PMID 31077668
- [Background] Arnold RW. Comparative AAPOS Validation of the Birefringent Amblyopia Screener with Isolated Small-Angle Strabismus. Clin Ophthalmol. 2020 Jan 31;14:325-329. doi: 10.2147/OPTH.S242335. eCollection 2020. PMID 32099317